CLINICAL TRIAL: NCT03045809
Title: Improving HIV Prevention and Sexual and Reproductive Health Care in High Risk Women in Rwanda Using Lessons Learnt From Previous Rinda Ubuzima Projects
Brief Title: Women's Improvement of Sexual Health (WISH) Demonstration Project
Acronym: WISH
Status: Completed | Type: Observational
Sponsor: Janneke van de Wijgert (Other)
Collaborators: Rinda Ubuzima, Rwanda (Unknown); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor-Investigator, Janneke van de Wijgert, Professor, University of Liverpool
Organization: University of Liverpool (Other)
Other Study IDs: UoL001208
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-07

CONDITIONS: Sexually Transmitted Disease; Bacterial Vaginosis; Vaginal Candidiasis; Urinary Tract Infections
Keywords: Syndromic management; Point of care testing
MeSH Terms: conditions — Sexually Transmitted Diseases; Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The only samples to be retained are two vaginal swabs per participant. DNA will be extracted for qPCR testing of select urogenital organisms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women at risk of urogenital infections: Adult women living in the city of Kigali who are at high risk of HIV/urogenital infections (defined as having had more than one sexual partner in the last 12 months OR having been treated for a sexually transmitted infection (STI) in the last 12 months) regardless of the presence of current urogenital symptoms. Women who are known to be HIV-positive and/or pregnant are not excluded. All eligible women will be offered urogenital infection point-of-care tests.
  Interventions: Diagnostic Test: Urogenital infection point-of-care tests

INTERVENTIONS:
Diagnostic Test: Urogenital infection point-of-care tests — Instead of syndromic management of symptomatic women, the study offers screening of high risk women regardless of symptoms using point-of-care tests for HIV, TV, and BV (all women), syphilis, NG, and CT (when risk score positive), and UTI (when symptomatic).

SUMMARY:
The current standard of care for urogenital infections in Rwanda is syndromic management. Many urogenital infections are asymptomatic and therefore completely missed, and the management of vaginal discharge syndrome is known to be suboptimal. The primary objective of this study is to evaluate whether it is feasible to improve urogenital infection care in high risk women in Kigali, Rwanda, using point of care (POC) diagnostic testing for HIV, Trichomonas vaginalis (TV), and bacterial vaginosis (BV) in all women; POC testing for Neisseria gonorrhoeae (NG), Chlamydia trachomatis (CT), and syphilis in pregnant women and women assessed to be at high risk for these infections using a risk scoring questionnaire; and management of vaginal candidiasis, urinary tract infection (UTI), genital ulcers/inguinal bubos, and lower abdominal pain in women reporting relevant symptoms. The secondary objectives of this study are 1) to evaluate the performance and 2) to obtain the opinions of Rwandan stakeholders.

DETAILED DESCRIPTION:
This is a cross-sectional study. The improved urogenital infection care services will be advertised to women in Kigali, Rwanda, targeting women with urogenital complaints as well as women without urogenital complaints who have had high risk behavior. The services will be available for free at the research clinic for the duration of the project. All consenting women who attend the research clinic during the study period will be offered:

1. Voluntary counselling and testing for HIV.
2. Urine pregnancy test if indicated and contraception counselling.
3. POC testing for UTI if UTI symptoms are present.
4. POC testing for TV and BV regardless of symptoms, and management of vaginal candidiasis based on symptom-reporting.
5. POC testing for syphilis and CT/NG if pregnant or considered at risk by risk scoring questionnaire.
6. Syndromic management of genital ulcers/inguinal bubos and lower abdominal pain.
7. Treatment and partner notification and treatment as appropriate, and referrals to antenatal, family planning, HIV and cervical cancer screening care.

Information about sociodemographics, risk behavior, sexual and reproductive health history and current urogenital symptoms will be collected during the clinic visit. Women can opt out of each service offered. Services will be delivered within one half day. However, women can choose to leave before all results are available, and be contacted by study staff when results are available, which is particularly relevant for women undergoing CT/NG POC testing (which takes about 90 minutes).

Vaginal swabs for storage will be taken from all consenting women (women can choose between self- or clinician-sampling) for additional research testing at the end of the study to allow for performance evaluation of the CT/NG, TV and BV POC tests.

Opinions of stakeholders will be gathered during workshops (one before and one after completion of the study) and in-depth interviews (IDIs).

ELIGIBILITY:
Inclusion Criteria:

* Female, at least 18 years old (no upper age limit)
* At high risk of HIV/STIs, defined as having had more than one sexual partner in the last 12 months OR having been treated for an STI in the last 12 months
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Already participated in this study before (each woman can only participate once)
* Participating in another health intervention study
* For any other reason as judged by the Principal Investigator (these reasons will be recorded)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women living in the city of Kigali who are at high risk of HIV/urogenital infections (defined as having had more than one sexual partner in the last 12 months OR having been treated for a sexually transmitted infection (STI) in the last 12 months) regardless of the presence of current urogenital symptoms. Women who are known to be HIV-positive and/or pregnant will not be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janneke van de Wijgert, MD PhD MPH, Principal Investigator — University of Liverpool
Locations (1):
- Rinda Ubuzima, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Undecided
The University of Liverpool and project investigators support open access but university-wide systems are not yet accessible and open access has not yet been negotiated with the Rwandan authorities.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At risk women regardless of symptoms were enrolled between 7-2016 and 3-2017. Recruitment activities were implemented by study staff with the help of community mobilizers. They organized recruitment meetings, and distributed flyers. Women were encouraged to refer their friends.
Pre-assignment Details: Women were eligible if aged 18 or older, and at risk of sexually transmitted infections (more than one sex partner and/or having been treated for at least one STI in the past year), with or without urogenital symptoms. HIV-positive and pregnant women were not excluded. Women were screened free of charge but did not receive a monetary reimbursement.
Groups:
- Women at Risk of Urogenital Infections.: All enrolled women attended one main study visit and underwent the same procedures. At the main study visit, participants underwent a face-to-face interview that included questions about current (incl. past two weeks) urogenital symptoms. This information was used to reconstruct WHO syndromic management diagnoses. Next, the WISH algorithms that incorporated point-of-care (POC) testing were implemented. All women were offered HIV, pregnancy, Trichomonas vaginalis (TV OSOM), and bacterial vaginosis (BV; vaginal pH; pH≥5.0 considered BV) POC testing. We only offered chlamydia/gonorrhea (CT/NG) GeneXpert testing to women who had a positive CT/NG risk score, and Determine syphilis POC testing to women who had a positive syphilis risk score. Vulvovaginal candidiasis (VVC) was treated presumptively. Treatment, partner notification, and/or referral procedures were offered as needed. Gold standard diagnoses were determined by testing samples from all women for BV, VVC, TV, NG, and CT by PCR.
Period: Overall Study
Arm/Group | Women at Risk of Urogenital Infections.
Started | 705
Attended an Additional Visit (if Needed) | 51 ((only if needed, for medical follow-up, to complete study procedures, or to report adverse events).)
Completed | 705
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 705 women who attended a main visit. Women were aged 18 or older, and at risk of sexually transmitted infections (more than one sex partner and/or having been treated for at least one STI in the past year), with or without urogenital symptoms. HIV-positive and pregnant women were not excluded.
Arm/Group | Women at Risk of Urogenital Infections.
Number analyzed (Participants) | 705
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 705
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 32.9 [18 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 705
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African (Rwandan) | 705
Region of Enrollment [Number; unit: participants]
  Rwanda | 705
Chlamydia trachomatis positive by gold standard test [Count of Participants; unit: Participants] | 60
Neisseria gonorrhoeae positive by gold standard test [Count of Participants; unit: Participants] | 50
Trichomonas vaginalis positive by gold standard test [Count of Participants; unit: Participants] | 111
Bacterial vaginosis positive by gold standard test [Count of Participants; unit: Participants] | 125

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Integrating Point-of-care Testing (Monitoring & Evaluation Indicators)
Description: Clinical monitoring and evaluation indicators: numbers of women with positive CT/NG or syphilis risk scores, number of pelvic exams done, etc (see row titles in the table)
Time Frame: Each participant was assessed at one main study visit, which lasted up to 4 hours.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Women at Risk of Urogenital Infections.
Number analyzed (Participants) | 705
Participants
  Had a positive CT/NG risk score | 396
  Had a positive syphilis risk score | 378
  Underwent a pelvic examination | 399
  Had any abnormality during the pelvic examination | 216
  Had at least one positive POCT result | 541
  Received all positive POCT results at main visit | 505
  Received inadequate treatment | 0
  Needed and received a referral | 79
  Had at least one partner requiring notification | 201
  Required at least one additional visit | 51

2. Primary Outcome: Feasibility of Integrating Point-of-care Testing (Client Satisfaction Surveys)
Description: Answers to questions about experiences with the procedures (client satisfaction survey).
Time Frame: Each client satisfaction survey was conducted at a main visit and lasted up to 30 min.
Population: A random selection of 107 enrolled women.
Measure: Count of Participants; unit: Participants
Arm/Group | Women at Risk of Urogenital Infections.
Number analyzed (Participants) | 107
Participants
  Felt welcome at study clinic | 107
  Thought medical services were of good quality | 107
  Thought counselling was of good quality | 107
  Thought visit duration was too long but worth it | 41
  Thought visit duration was too long and not worth | 0
  Willing to be tested in future even if asymptomati | 100
  Willing to pay for services in future: number analyzed (Participants) | 106
  Willing to pay for services in future | 95

3. Primary Outcome: Performance of Syndromic Management With or Without Integration of Point-of-care Tests
Description: With performance we mean sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). We determined the number of women who would have received treatment for BV, VVC, TV, NG, and/or CT in the following situations: 1) if we would have followed the WHO syndromic management algorithms for vaginal discharge and lower abdominal pain; and 2) based on the POCT-based WISH algorithms (this is what we did in real life during the study), and compared each of these with gold standard infection-specific diagnoses. The results of the first comparison are reported in the first column and results of the second comparison in the second column.
Time Frame: Each participant was assessed at one main study visit, which lasted up to 4 hours.
Population: Gold standard results availability ranged between 690 to 705 per separate outcome. For CT and NG, results were available for all 705 participants. For BV, VVC, and TV, 690 results were available (15 PCR results were invalid).
Measure: Number (95% Confidence Interval); unit: % (sensitivity/specificity/PPV/NPV)
Groups:
- WHO Syndromic Management (Entire Study Population): Syndromic management vs gold standard.
  With performance we mean sensitivity, specificity, positive predictive value, and negative predictive value. We determined the number of women who would have received treatment for BV, VVC, TV, NG, and/or CT if we would have followed the WHO syndromic management algorithms for vaginal discharge and lower abdominal pain; and compared this with gold standard infection-specific diagnoses.
- WISH (Entire Study Population): WISH POCT vs gold standard
  With performance we mean sensitivity, specificity, positive predictive value, and negative predictive value. We determined the number of women who had received treatment for BV, VVC, TV, NG, and/or CT based on the POCT-based WISH algorithms (this is what we did in real life during the study), and compared this with gold standard infection-specific diagnoses.
Arm/Group | WHO Syndromic Management (Entire Study Population) | WISH (Entire Study Population)
Number analyzed (Participants) | 705 | 705
% (sensitivity/specificity/PPV/NPV)
  Chlamydia sensitivity | 58.3 [45.5 to 70.2] | 71.7 [58.3 to 81.7]
  Chlamydia specificity | 44.7 [40.8 to 48.5] | 100 [100 to 100]
  Chlamydia PPV | 8.9 [6.5 to 12.1] | 100 [100 to 100]
  Chlamydia NPV | 92 [88.4 to 94.6] | 97.4 [95.9 to 98.4]
  Gonorrhea sensitivity | 66.0 [51.8 to 77.8] | 76.0 [62.2 to 85.9]
  Gonorrhea specificity | 45.2 [41.4 to 49.0] | 100 [100 to 100]
  Gonorrhea PPV | 8.4 [6.0 to 11.6] | 100 [100 to 100]
  Gonorrhea NPV | 94.6 [91.4 to 96.6] | 98.2 [96.9 to 99.0]
  Trichomonas vaginalis sensitivity: number analyzed (Participants) | 690 | 690
  Trichomonas vaginalis sensitivity | 60.4 [50.9 to 69.1] | 68.5 [59.2 to 76.5]
  Trichomonas vaginalis specificity: number analyzed (Participants) | 690 | 690
  Trichomonas vaginalis specificity | 45.6 [41.6 to 49.7] | 97.4 [95.7 to 98.4]
  Trichomonas vaginalis PPV: number analyzed (Participants) | 690 | 690
  Trichomonas vaginalis PPV | 17.5 [14.0 to 21.7] | 83.5 [74.4 to 89.8]
  Trichomonas vaginalis NPV: number analyzed (Participants) | 690 | 690
  Trichomonas vaginalis NPV | 85.7 [81.3 to 89.2] | 94.2 [92.0 to 95.8]
  Bacterial vaginosis sensitivity: number analyzed (Participants) | 690 | 690
  Bacterial vaginosis sensitivity | 61.6 [52.7 to 69.7] | 95.2 [89.7 to 97.8]
  Bacterial vaginosis specificity: number analyzed (Participants) | 690 | 690
  Bacterial vaginosis specificity | 46.0 [41.9 to 50.2] | 41.2 [37.2 to 45.4]
  Bacterial vaginosis PPV: number analyzed (Participants) | 690 | 690
  Bacterial vaginosis PPV | 20.2 [16.4 to 24.5] | 26.4 [22.5 to 30.7]
  Bacterial vaginosis NPV: number analyzed (Participants) | 690 | 690
  Bacterial vaginosis NPV | 84.4 [79.9 to 88.1] | 97.5 [94.5 to 98.9]
  Vulvovaginal candidiasis sensitivity: number analyzed (Participants) | 690 | 690
  Vulvovaginal candidiasis sensitivity | 74.6 [61.9 to 84.1] | 64.4 [51.4 to 75.6]
  Vulvovaginal candidiasis specificity: number analyzed (Participants) | 690 | 690
  Vulvovaginal candidiasis specificity | 50.6 [46.6 to 54.5] | 69.4 [65.7 to 72.9]
  Vulvovaginal candidiasis PPV: number analyzed (Participants) | 690 | 690
  Vulvovaginal candidiasis PPV | 12.4 [9.3 to 16.2] | 16.5 [12.2 to 21.8]
  Vulvovaginal candidiasis NPV: number analyzed (Participants) | 690 | 690
  Vulvovaginal candidiasis NPV | 95.5 [92.7 to 97.3] | 95.4 [93.1 to 97.0]

ADVERSE EVENTS:
Time Frame: Each participant was assessed at one main study visit, which lasted up to 4 hours.
Arm/Group | Women at Risk of Urogenital Infections.
All-Cause Mortality (participants affected / at risk) | 0/705
Serious Adverse Events (participants affected / at risk) | 0/705
Other Adverse Events (participants affected / at risk) | 2/705
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women at Risk of Urogenital Infections. (N=705)
Allergic reaction to metronidazole (Skin and subcutaneous tissue disorders) | 2 (2) — Allergic reaction to metronidazole; also included nausea, vomiting.

LIMITATIONS AND CAVEATS:
The study was implemented in a high prevalence population by experienced staff. Additional studies are required in low prevalence settings and in public primary care clinics. Our recruitment strategies mostly attracted women with symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03045809/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT03045809/SAP_001.pdf